CLINICAL TRIAL: NCT01197365
Title: Double-blind Randomized Controlled Study for the Evaluation of Nutritional Outcomes of a Cow's Milk Based Infant Formula Containing Galacto-oligosaccharides, Beta-palmitate and Acidified Milk
Brief Title: Safety and Efficacy of an Infant Formula Supplemented With Galacto-oligosaccharides, Beta-palmitate and Acidified Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinz Italia SpA (Industry)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Centro di Immunità e Nutrizione - Università degli Studi di Pavia (Prof.ssa Annamaria Castellazzi) (Unknown); Advanced Analytical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PLA-LENI-09
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Formula Feeding of Healthy Full Term Infants
Keywords: Acidified milk; Beta-palmitate; Bifidobacteria; Infant formula; Galacto-oligosaccharides; Growth; Infants; Prebiotics
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- STUDY GROUP (Experimental): Infant formula supplemented with functional ingredients (galacto-oligosaccharides, beta-palmitate, acidified milk.
  Infant formula with functional ingredients is in compliance with Directive 2006/141/CE on infant formulae and follow-on formulae
  Interventions: Other: Infant formula with GOS, beta-palmitate, acidified milk
- CONTROL GROUP (Other): Standard infant formula, in compliance with Directive 2006/141/CE on infant formulae and follow-on formulae, without functional ingredients
  Interventions: Other: Standard infant formula without functional ingredients

INTERVENTIONS:
Other: Infant formula with GOS, beta-palmitate, acidified milk — Infant formula supplemented with functional ingredients (galacto-oligosaccharides, beta-palmitate, acidified milk.
  Infant formula with functional ingredients is in compliance with Directive 2006/141/CE on infant formulae and follow-on formulae
  Arms: STUDY GROUP
Other: Standard infant formula without functional ingredients — Standard infant formula, in compliance with Directive 2006/141/CE on infant formulae and follow-on formulae, without functional ingredients
  Arms: CONTROL GROUP

SUMMARY:
The purpose of this study is to determine the safety and efficacy of an infant formula supplemented with galacto-oligosaccharides (GOS), beta-palmitate and acidified milk in improving the gastrointestinal health and immune response in healthy term infants.

DETAILED DESCRIPTION:
Infant formulae are the only alternatives to breast milk for infants when, for whatever reason, human milk becomes unavailable.

New-generation infant formulae contain functional ingredients able to mimic some benefits of human milk.

The study formula is supplemented with galacto-oligosaccharides, which favor intestinal positive microflora growth, beta-palmitate, enhancing fat and calcium absorption and softer stool formation, and acidified milk which contributes to immune system maturation.

The aim of this study is to verify the safety of the study formula in healthy term infants and to deepen the efficacy of the functional ingredient blend in term of prebiotic effect, gastrointestinal tolerance and immune response improvement.

ELIGIBILITY:
Inclusion Criteria:

* Infants of both sexes born to natural or cesarean delivery
* Gestational age between 37 and 42 completed weeks
* Birth weight between 10th and 90th percentile of birth weight for gestational age, according to the North-Italian growth charts
* Single birth
* Caucasian parents
* Infants being exclusively formula-fed by the 21st day of life

Exclusion Criteria:

* Infants with genetic and/or congenital diseases
* Infants receiving antibiotic therapy
* Infants with neonatal diseases requiring hospitalisation for longer than 7 days
* Infants at risk for atopy and/or having familial history for atopy
* Mothers with metabolic or chronic diseases
* Infant selected for another clinical study
* Parents refusing to sign a written informed consent

Max Age: 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2010-08; Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The nutritional safety of the study formula is evaluated through measure of anthropometric parameters and record of gastrointestinal symptoms | Anthropometric parameters: at birth, at enrolment, after 60 and 135 days of life. Gastrointestinal symptoms: recorded daily in the infant's diary.
  Anthropometric parameters: body weight, recumbent length and head circumference change. Gastrointestinal symptoms: diarrhea, constipation, stool frequency and consistency, bowel cramps, abdominal distension, intestinal gas.

SECONDARY OUTCOMES:
Immune-modulatory activity | At enrolment, after 60 and 135 days of life
  Quantification of salivary IgA
Prebiotic effect | At enrolment and after 135 days of life
  Microbiological analysis of feces

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Stronati, Prof., Principal Investigator — FONDAZIONE IRCCS POLICLINICO "SAN MATTEO" - STRUTTURA COMPLESSA DI NEONATOLOGIA, PATOLOGIA NEONATALE E TERAPIA INTENSIVA
Locations (1):
- Fondazione Irccs Policlinico "San Matteo" - Struttura Complessa Di Neonatologia, Patologia Neonatale E Terapia Intensiva, Pavia, PV, Italy

REFERENCES:
- [Background] Aggett PJ, Agostini C, Goulet O, Hernell O, Koletzko B, Lafeber HL, Michaelsen KF, Rigo J, Weaver LT; European Society of Pediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN) Committee on Nutrition. The nutritional and safety assessment of breast milk substitutes and other dietary products for infants: a commentary by the ESPGHAN Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2001 Mar;32(3):256-8. doi: 10.1097/00005176-200103000-00004. No abstract available. PMID 11345171
- [Background] Carver JD. Advances in nutritional modifications of infant formulas. Am J Clin Nutr. 2003 Jun;77(6):1550S-1554S. doi: 10.1093/ajcn/77.6.1550S. PMID 12812153
- [Background] Agostoni C, Axelsson I, Goulet O, Koletzko B, Michaelsen KF, Puntis JW, Rigo J, Shamir R, Szajewska H, Turck D; ESPGHAN Committee on Nutrition. Prebiotic oligosaccharides in dietetic products for infants: a commentary by the ESPGHAN Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2004 Nov;39(5):465-73. doi: 10.1097/00005176-200411000-00003. PMID 15572882
- [Background] Brunser O, Araya M, Espinoza J, Guesry PR, Secretin MC, Pacheco I. Effect of an acidified milk on diarrhoea and the carrier state in infants of low socio-economic stratum. Acta Paediatr Scand. 1989 Mar;78(2):259-64. doi: 10.1111/j.1651-2227.1989.tb11066.x. PMID 2929349
- [Background] Mullie C, Yazourh A, Thibault H, Odou MF, Singer E, Kalach N, Kremp O, Romond MB. Increased poliovirus-specific intestinal antibody response coincides with promotion of Bifidobacterium longum-infantis and Bifidobacterium breve in infants: a randomized, double-blind, placebo-controlled trial. Pediatr Res. 2004 Nov;56(5):791-5. doi: 10.1203/01.PDR.0000141955.47550.A0. Epub 2004 Sep 3. PMID 15347767
- [Background] Thibault H, Aubert-Jacquin C, Goulet O. Effects of long-term consumption of a fermented infant formula (with Bifidobacterium breve c50 and Streptococcus thermophilus 065) on acute diarrhea in healthy infants. J Pediatr Gastroenterol Nutr. 2004 Aug;39(2):147-52. doi: 10.1097/00005176-200408000-00004. PMID 15269618
- [Background] Lucas A, St James-Roberts I. Crying, fussing and colic behaviour in breast- and bottle-fed infants. Early Hum Dev. 1998 Nov;53(1):9-18. doi: 10.1016/s0378-3782(98)00032-2. PMID 10193923
- [Background] Quinlan PT, Lockton S, Irwin J, Lucas AL. The relationship between stool hardness and stool composition in breast- and formula-fed infants. J Pediatr Gastroenterol Nutr. 1995 Jan;20(1):81-90. doi: 10.1097/00005176-199501000-00014. PMID 7884622
- [Background] Billeaud C, Guillet J, Sandler B. Gastric emptying in infants with or without gastro-oesophageal reflux according to the type of milk. Eur J Clin Nutr. 1990 Aug;44(8):577-83. PMID 2209513
- [Background] Carnielli VP, Luijendijk IH, van Goudoever JB, Sulkers EJ, Boerlage AA, Degenhart HJ, Sauer PJ. Feeding premature newborn infants palmitic acid in amounts and stereoisomeric position similar to that of human milk: effects on fat and mineral balance. Am J Clin Nutr. 1995 May;61(5):1037-42. doi: 10.1093/ajcn/61.4.1037. PMID 7733025
- [Background] Carnielli VP, Luijendijk IH, van Beek RH, Boerma GJ, Degenhart HJ, Sauer PJ. Effect of dietary triacylglycerol fatty acid positional distribution on plasma lipid classes and their fatty acid composition in preterm infants. Am J Clin Nutr. 1995 Oct;62(4):776-81. doi: 10.1093/ajcn/62.4.776. PMID 7572708
- [Background] Carnielli VP, Luijendijk IH, Van Goudoever JB, Sulkers EJ, Boerlage AA, Degenhart HJ, Sauer PJ. Structural position and amount of palmitic acid in infant formulas: effects on fat, fatty acid, and mineral balance. J Pediatr Gastroenterol Nutr. 1996 Dec;23(5):553-60. doi: 10.1097/00005176-199612000-00007. PMID 8985844
- [Background] Lucas A, Quinlan P, Abrams S, Ryan S, Meah S, Lucas PJ. Randomised controlled trial of a synthetic triglyceride milk formula for preterm infants. Arch Dis Child Fetal Neonatal Ed. 1997 Nov;77(3):F178-84. doi: 10.1136/fn.77.3.f178. PMID 9462186
- [Background] Kennedy K, Fewtrell MS, Morley R, Abbott R, Quinlan PT, Wells JC, Bindels JG, Lucas A. Double-blind, randomized trial of a synthetic triacylglycerol in formula-fed term infants: effects on stool biochemistry, stool characteristics, and bone mineralization. Am J Clin Nutr. 1999 Nov;70(5):920-7. doi: 10.1093/ajcn/70.5.920. PMID 10539755
- [Background] Lopez-Lopez A, Castellote-Bargallo AI, Campoy-Folgoso C, Rivero-Urgel M, Tormo-Carnice R, Infante-Pina D, Lopez-Sabater MC. The influence of dietary palmitic acid triacylglyceride position on the fatty acid, calcium and magnesium contents of at term newborn faeces. Early Hum Dev. 2001 Nov;65 Suppl:S83-94. doi: 10.1016/s0378-3782(01)00210-9. PMID 11755039
- [Background] Nelson CM, Innis SM. Plasma lipoprotein fatty acids are altered by the positional distribution of fatty acids in infant formula triacylglycerols and human milk. Am J Clin Nutr. 1999 Jul;70(1):62-9. doi: 10.1093/ajcn/70.1.62. PMID 10393140
- [Background] Mackie RI, Sghir A, Gaskins HR. Developmental microbial ecology of the neonatal gastrointestinal tract. Am J Clin Nutr. 1999 May;69(5):1035S-1045S. doi: 10.1093/ajcn/69.5.1035s. PMID 10232646
- [Background] Zoppi G, Cinquetti M, Luciano A, Benini A, Muner A, Bertazzoni Minelli E. The intestinal ecosystem in chronic functional constipation. Acta Paediatr. 1998 Aug;87(8):836-41. doi: 10.1080/080352598750013590. PMID 9736230
- [Background] Mountzouris KC, McCartney AL, Gibson GR. Intestinal microflora of human infants and current trends for its nutritional modulation. Br J Nutr. 2002 May;87(5):405-20. doi: 10.1079/BJNBJN2002563. PMID 12010580
- [Background] Savino F, Cresi F, Pautasso S, Palumeri E, Tullio V, Roana J, Silvestro L, Oggero R. Intestinal microflora in breastfed colicky and non-colicky infants. Acta Paediatr. 2004 Jun;93(6):825-9. PMID 15244234
- [Background] Tlaskalova-Hogenova H, Stepankova R, Hudcovic T, Tuckova L, Cukrowska B, Lodinova-Zadnikova R, Kozakova H, Rossmann P, Bartova J, Sokol D, Funda DP, Borovska D, Rehakova Z, Sinkora J, Hofman J, Drastich P, Kokesova A. Commensal bacteria (normal microflora), mucosal immunity and chronic inflammatory and autoimmune diseases. Immunol Lett. 2004 May 15;93(2-3):97-108. doi: 10.1016/j.imlet.2004.02.005. PMID 15158604
- [Background] Ben XM, Li J, Feng ZT, Shi SY, Lu YD, Chen R, Zhou XY. Low level of galacto-oligosaccharide in infant formula stimulates growth of intestinal Bifidobacteria and Lactobacilli. World J Gastroenterol. 2008 Nov 14;14(42):6564-8. doi: 10.3748/wjg.14.6564. PMID 19030213
- [Background] Fanaro S, Marten B, Bagna R, Vigi V, Fabris C, Pena-Quintana L, Arguelles F, Scholz-Ahrens KE, Sawatzki G, Zelenka R, Schrezenmeir J, de Vrese M, Bertino E. Galacto-oligosaccharides are bifidogenic and safe at weaning: a double-blind randomized multicenter study. J Pediatr Gastroenterol Nutr. 2009 Jan;48(1):82-8. doi: 10.1097/MPG.0b013e31817b6dd2. PMID 19172129
- [Background] Ben XM, Zhou XY, Zhao WH, Yu WL, Pan W, Zhang WL, Wu SM, Van Beusekom CM, Schaafsma A. Supplementation of milk formula with galacto-oligosaccharides improves intestinal micro-flora and fermentation in term infants. Chin Med J (Engl). 2004 Jun;117(6):927-31. PMID 15198901
- [Background] World Health Organization. Nutrient adequacy of exclusive breastfeeding for the term infant during the first six months of life. Geneva, 2002.
- [Derived] Civardi E, Garofoli F, Longo S, Mongini ME, Grenci B, Mazzucchelli I, Angelini M, Castellazzi A, Fasano F, Grinzato A, Fanos V, Budelli A, Stronati M. Safety, growth, and support to healthy gut microbiota by an infant formula enriched with functional compounds. Clin Nutr. 2017 Feb;36(1):238-245. doi: 10.1016/j.clnu.2015.11.006. Epub 2015 Nov 27. PMID 26718667